CLINICAL TRIAL: NCT05935540
Title: Effects of a Structured, Family-supported, Patient-centred Advance Care Planning for End-of-life Decision Among Palliative Care Patients and Their Family Members: a Randomized Controlled Trial
Brief Title: ACP-Family Programme for Palliative Care Patients and Their Family Member
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shatin Hospital (Other); United Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ACP2023
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-08

CONDITIONS: Palliative Care
Keywords: Advance care planning; palliative care; family; decision making

STUDY DESIGN:
Intervention Model Description: A parallel, 2-armed RCT with follow-ups at 6 and 12 months
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACP-Family (Experimental): It is a ACP discussion intervention consisting of two sessions (45-60 mins) and to be delivered within one month in a face-to-face format as long as the patient is still in the hospital by a trained ACP facilitator.
  Interventions: Other: ACP-Family
- ACP-UC (No Intervention): Usual care that is available to all palliative care patients in the hospital.

INTERVENTIONS:
Other: ACP-Family — It consists of two sessions (45-60 mins) to be delivered within one month in a face-to-face format as long as the patient is still in the hospital. The treatment will be continued in the patient's home if he/she is discharged before the two sessions are completed.
  The treatment will cover five elements in ACP, namely (1) patients' understanding of their illness, (2) patients' values and beliefs underpinning care preferences, (3) possible health conditions in the future, (4) introducing the idea of AD and its arrangement, and (5) construction of the role of substituted decision maker. A 3-min video on end-of-life treatment options will be shown to help patients and family members to clearly understand the related topic. However, there will be no restriction on the order of the five topics to be discussed during the intervention.
  Other Names: Structured, family-supported, patient-centred ACP
  Arms: ACP-Family

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a structured, family-supported, patient-centred advance care planning (ACP) in palliative care patients and their family members. The main question it aims to answer is: • the effectiveness of the ACP intervention on promoting end-of-life decision making and psychological outcomes in patients and family members. Participants will be assigned to either the ACP-Family group (ACP-Family) to receive a structured, family-supported, patient-centred ACP intervention or usual palliative care (ACP-UC) at the hospital. Researchers will compare the ACP-Family and ACP-UC groups to see if the ACP-Family group will produce better outcomes than the ACP-UC group.

DETAILED DESCRIPTION:
This is a two-arm parallel randomized controlled trial with follow-ups at 6 and 12 months, aiming to examine the effectiveness of a structured, family-supported, patient-centred ACP programme for adult palliative care patients and their families.

This study will randomize 170 palliative care patients and their family members to the structured, family-supported, patient-centred ACP programme (ACP-Family) or ACP service under usual care (ACP-UC). Within one month, they will receive two 60-90 minute sessions of the family-supported, patient-centred ACP programme covering five elements in ACP discussions delivered by a trained ACP facilitator; or usual care provided by the respective hospital. All discussion sessions in the ACP group will be recorded for quality checking.

It is hypothesized that, as compare to ACP-UC, the ACP-Family group will significantly improve EOL decision making outcomes including (i) prediction accuracy of patient's treatment preferences between palliative care patients and their family members, (ii) new ACP documentation in palliative care patients, and (iii) family-reported patient's EOL care preferences was respected for deceased patients; and 2. psychological outcomes including family member's decision-making confidence, anxiety, depression, and quality of communication regarding EOL, and patient's decisional conflict, and perceived quality of communication regarding EOL.

In addition, 3. we also explore the potential moderating effect of type of hospital setting on the effectiveness of the ACP-Family on these patient and family outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* aged ≥ 18,
* receiving palliative care at the study hospitals,
* able to communicate in Cantonese, and
* cognitively intact (Abbreviated Mental Test (AMT) score ≥ 7)13 at the time of recruitment

Family member:

* aged≥ 18
* able to communicate in Cantonese, and
* nominated by the patient who is likely to make substituted decisions for the patient in future health care issues.

Exclusion Criteria:

* are engaging in ACP discussion with healthcare professionals in the hospital at the time of recruitment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Family's prediction accuracy of patient's treatment preferences | 6 months
  Patients and family members will be asked independently to indicate patient's preferences regarding three life-sustaining treatments (cardiopulmonary resuscitation, mechanical ventilator and tube feeding) based on three options (want to attempt, refuse or uncertain) in two hypothetical EOL scenarios (being terminally ill and in persistent vegetative state or a state of irreversible coma). An accuracy score will be calculated by summing the number of treatment decisions for which responses from the patient and family member are identical, and then dividing by the total number of decisions (n = 6), all equally weighted.

SECONDARY OUTCOMES:
Family's prediction accuracy of patient's treatment preferences | 12 months
  Patients and family members will be asked independently to indicate patient's preferences regarding three life-sustaining treatments (cardiopulmonary resuscitation, mechanical ventilator and tube feeding) based on three options (want to attempt, refuse or uncertain) in two hypothetical EOL scenarios (being terminally ill and in persistent vegetative state or a state of irreversible coma). An accuracy score will be calculated by summing the number of treatment decisions for which responses from the patient and family member are identical, and then dividing by the total number of decisions (n = 6), all equally weighted.
New ACP documentation | 6 and 12 months
  Advance directives will be retrieved from medical record or ACP discussion recorded reported by the patients or family member. A composite variable of any ACP documentation (forms and/or discussion) will be created.
Family-reported perception of whether the patient's EOL care preference was respected | 6 and 12 months
  For deceased patients, their family members will be asked to respond to two items (whether EOL wishes were discussed and whether they were met) and a binary variable will be generated.
Patient's decisional conflict | 6 and 12 months
  Patient's decisional conflict in making decisions related to future care will be measured by the SURE test scale. Patients will be asked to rate their future care on four items using a Yes/No format.
Quality of communication | 6 and 12 months
  Patient-healthcare provider and family-healthcare provider quality of communication about EOL care will be measured using the corresponding subscale of the validated Quality of Communication Questionnaire. Patients and family members will be asked to rate how good their physician is at each of the 7 communication skills about EOL discussion.
Family's decision-making confidence | 6 and 12 months
  Family's decision-making confidence in EOL decision making for their patients will be measured by the 5-item Decision Making Confidence Scale. Family members will be asked to indicate their level of comfort in the surrogate role on a 5-point Likert scale.
Family's anxiety and depression | 6 and 12 months
  Family's anxiety and depression will be assessed by the widely used 14-item Hospital Anxiety and Depression Scale (HADS). The HADS consists of two subscales: anxiety (7 items) and depression (7 items) with scores range 0-21
Satisfaction to the intervention | 6 months
  Patients and family members in the ACP-Family arm will be asked to rate their satisfaction about the discussion, the video shown, the ACP facilitator and the involvement of the family member (for patient only) using one item on a 0-10 VAS scale separately

CONTACTS AND LOCATIONS:
Overall Officials: Doris YP Leung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - Bradbury Hospice, Hong Kong
  - Shatin Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not readily shared because permission to use the data by other researchers has to seek approval from the ethical committee. Requests to access IPD should be directed to PI for further consideration and seeking approval from ethical committee.

REFERENCES:
- [Derived] Leung DYP, Chung JOK, Chan HYL, Lo RSK, Li K, Lam PT, Ng NHY. Effects of a structured, family-supported, and patient-centred advance care planning on end-of-life decision making among palliative care patients and their family members: protocol of a randomised controlled trial. BMC Palliat Care. 2024 Nov 7;23(1):257. doi: 10.1186/s12904-024-01588-z. PMID 39511666